CLINICAL TRIAL: NCT00446290
Title: A Phase I Study of Docetaxel, Capecitabine and Oxaliplatin (DXO) in Patients With Advanced Stomach Cancer
Brief Title: Study of Docetaxel, Capecitabine and Oxaliplatin in Advanced Stomach Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Yoon-Koo Kang, Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMC0609
Record Dates: First submitted 2007-03-09; First posted 2007-03-12 (Estimated); Results first posted 2015-07-28 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Stomach Cancer
Keywords: To determine maximal tolerated dose of DXO regimen
MeSH Terms: conditions — Stomach Neoplasms | interventions — Docetaxel; Capecitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Docetaxel, Capecitabine and Oxaliplatin (Experimental)
  Interventions: Drug: Docetaxel, Capecitabine and Oxaliplatin

INTERVENTIONS:
Drug: Docetaxel, Capecitabine and Oxaliplatin

SUMMARY:
Considering synergism between docetaxel (D), capecitabine (X), and oxaliplatin (O) and favourable toxicity profile of oxaliplatin over cisplatin, it is to be expected that combination of docetaxel, capecitabine, and oxaliplatin (DXO) will be more effective than other regimens and feasible in advanced gastric cancer. DXO regimen can be also easily administered on out-patient setting. However, so far, DXO combination has not been tried in advanced gastric cancer. The investigators will determine maximum tolerated dose of DXO regimen in this phase I study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed unresectable or metastatic advanced gastric adenocarcinoma
* Completion of adjuvant chemotherapy 6 months before the study, or no previous chemotherapy (But, patients who received docetaxel, capecitabine, or oxaliplatin as adjuvant chemotherapy should be excluded.)
* Age 18 to 70 years old
* Eastern Cooperative Oncology Group performance status 0~2
* Adequate bone marrow function: white blood cell counts >4,000/µL, absolute neutrophil count >2,000/µL, and platelets>100,000/µL
* Adequate renal function: creatinine < 1 x upper normal limit (UNL) or creatinine clearance 60ml/min
* Adequate hepatic function: bilirubin < 1.5 x UNL, aspartate aminotransferase (AST)/alanine aminotransferase (ALT) levels < 2.5 x UNL, and alkaline phosphatase < 5 x UNL (except in case of bone metastasis without any liver disease)
* Given written informed consent prior to study-specific screening procedures, with the understanding that the patient has the right to withdraw from the study at any time, without prejudice

Exclusion Criteria:

* Contraindication to any drug contained in the chemotherapy regimen
* Other tumor type than adenocarcinoma
* Presence or history of central nervous system (CNS) metastasis
* Gastric outlet or bowel obstruction
* Evidence of serious gastrointestinal bleeding
* Peripheral neuropathy > grade 1
* History of significant neurologic or psychiatric disorders
* History of another malignancy within the last five years except cured basal cell carcinoma of skin and cured carcinoma in-situ of uterine cervix
* Pregnant or lactating women, women of childbearing potential not employing adequate contraception. Postmenopausal women must have been amenorrheic for at least 12 months to be considered of non-childbearing potential
* Sexually active males and females (of childbearing potential) unwilling to practice conception during the study
* Clinically significant cardiac disease (e.g. severe non-compensated hypertension, non-compensated heart failure, dilated cardiomyopathy, and coronary heart disease with ST segment depression in electrocardiogram) or myocardial infarction within the last 6 months
* Serious pulmonary conditions/illness (e.g. chronic lung disease with hypoxemia)
* Serious metabolic disease such as severe non-compensated diabetes mellitus
* Serious uncontrolled intercurrent infections, or other serious uncontrolled concomitant disease
* Positive serology for the human immunodeficiency virus (HIV)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2006-03; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yoon-Koo Kang, MD, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Groups:
- DXO Arm: Docetaxel, capecitabine and oxaliplatin
  Dose level Docetaxel(mg/m2) Capecitabine(mg/m2, twice daily) Oxaliplatin(mg/m2)
  1. 45 800 100
  2. 60 800 100
  3. 60 1,000 100
  4. 60 800 130
  5. 60 1,000 130
Period: Overall Study
Arm/Group | DXO Arm
Started | 22
Completed | 22
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- DXP Arm: Docetaxel, capecitabine and oxaliplatin
Arm/Group | DXP Arm
Number analyzed (Participants) | 21
Age, Customized [Median (Full Range); unit: years] | 50 [21 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 21
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 21

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With DLTs
Description: Dose limiting toxicity (DLTs) was determined during the Wrst two cycles of treat- ment. The definitions of DLTs were as follows: (1) grade 4 neutropenia lasting for more than 5 days, or grade 3/4 neu- tropenia with fever; (2) grade 4 thrombocytopenia; (3) any other grade 3 non-hematological toxicity (excluding alope- cia); or (4) treatment delay of more than 2 weeks following the time of planned treatment. Maximal tolerated dose was defined as that the DLTs were observed in two or more patients from a cohort of two to six patients
Time Frame: 2 years
Population: All patients who were initially enrolled in dose escalation scheme.
Measure: Number; unit: participants
Groups:
- DXO Arm: Docetaxel, capecitabine and oxaliplatin
Arm/Group | DXO Arm
Number analyzed (Participants) | 15
participants | 3

ADVERSE EVENTS:
Time Frame: 6 months after completion of study treatment. If patients received another treatment, further evaluation was not done.
Arm/Group | DXO Arm
Serious Adverse Events (participants affected / at risk) | 7/21
Other Adverse Events (participants affected / at risk) | 12/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DXO Arm (N=21)
Febrile neutropenia (Infections and infestations) | 6
Diarrhea (Gastrointestinal disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DXO Arm (N=22)
Anemia (Blood and lymphatic system disorders) | 11
Leukopenia (Blood and lymphatic system disorders) | 10
Neutropenia (Blood and lymphatic system disorders) | 11
Thrombocytopenia (Blood and lymphatic system disorders) | 8
Febrile neutropenia (Infections and infestations) | 3
Asthenia (General disorders) | 12
Nausea (Gastrointestinal disorders) | 10
Vomiting (Gastrointestinal disorders) | 5
Stomatitis (Gastrointestinal disorders) | 7
Diarrhea (Gastrointestinal disorders) | 8
Nail toxicity (Skin and subcutaneous tissue disorders) | 9
Neuropathy (Nervous system disorders) | 8
Hand-foot syndrome (Skin and subcutaneous tissue disorders) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No